CLINICAL TRIAL: NCT00999661
Title: A Study of Clinical Outcomes of the REALIZE Adjustable Gastric Band-C at 2 Years in a US Patient Population of Morbidly Obese Patients
Brief Title: A Study of Clinical Outcomes of the REALIZE Adjustable Gastric Band-C
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-09-0007
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the results patients are obtaining with the Realize™ Adjustable Gastric Band-C during the first 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Received an implant with the Realize Band-C according to the following indications for use:

   1. Body Mass Index (BMI) of at least 40 kg/m2, or a BMI of at least 35 kg/m2 with one or more co-morbid conditions.
   2. Male and female adult patients (adult is defined as 18 years of age or older)
   3. Failed more conservative weight-reduction alternatives, such as supervised diet, exercise, and behavior modification programs.
2. Able to comprehend, follow, and give signed informed consent.

Exclusion Criteria:

1. Inflammatory diseases of the gastrointestinal tract, including severe intractable esophagitis, gastric ulceration or duodenal ulceration, or specific inflammation such as Crohn's disease;
2. Severe cardiopulmonary disease or other serious organic disease;
3. Upper gastrointestinal bleeding conditions such as esophageal or gastric varices or intestinal telangiectases;
4. Portal hypertension;
5. Anomalies of the gastrointestinal tract such as atresia or stenosis;
6. Cirrhosis of the liver;
7. Chronic pancreatitis;
8. Localized or systemic infection;
9. On chronic, long-term systemic steroid treatment or systemic steroids within 15 days of surgery;
10. Unable or unwilling to comply with dietary restrictions required by this procedure;
11. Known allergy to materials contained in the gastric band or its Injection Port;
12. Women who are pregnant;
13. Women at childbearing potential planning to get pregnant within 2 years or not using acceptable methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At each participating center (after the initial 10 cases), all consecutively implanted patients, will be considered for the study.
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Los Angeles, California
  - Celebration, Florida
  - Joliet, Illinois
  - Holland, Michigan
  - Patchogue, New York
  - Charlotte, North Carolina
  - Houston, Texas

REFERENCES:
- [Result] Cunneen SA, Brathwaite CE, Joyce C, Gersin K, Kim K, Schram JL, Wilson EB, Schwiers M, Gutierrez M. Clinical outcomes of the Realize Adjustable Gastric Band-C at 2 years in a United States population. Surg Obes Relat Dis. 2013 Nov-Dec;9(6):885-93. doi: 10.1016/j.soard.2013.02.009. Epub 2013 Mar 14. PMID 23642493
- [Result] Cunneen SA, Brathwaite CE, Joyce C, Gersin K, Kim K, Schram JL, Wilson EB, Rodriguez CE, Gutierrez M. Clinical outcomes of the REALIZE adjustable gastric band-C at one year in a U.S. population. Surg Obes Relat Dis. 2012 May-Jun;8(3):288-95. doi: 10.1016/j.soard.2011.05.004. Epub 2011 May 20. PMID 21775219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment began in November, 2009 at 7 surgical centers in the United States.
Pre-assignment Details: This was a longitudinal, single arm, observational, non-comparative study of clinical outcomes. Subjects were asked to consent to data collection to the study parameters from their study records.
Groups:
- Realize Adjustable Gastric Band-C: All subjects implanted with the Realize Gastric Band-C.
Period: Overall Study
Arm/Group | Realize Adjustable Gastric Band-C
Started | 231
Completed | 161
Not Completed | 70
Not completed — Lost to Follow-up | 59
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Not meeting eligibility criteria | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population defined as all subjects implanted with the Realize Gastric Band-C who signed informed consent.
Arm/Group | Realize Adjustable Gastric Band-C
Number analyzed (Participants) | 231
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 214
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 231

OUTCOME MEASURES:

1. Primary Outcome: Percent Excess Weight Change From Baseline to 24 Months
Description: Percent excess weight change from baseline to 24 months was calculated as (the baseline weight minus the weight at 24 months) divided by the (baseline weight minus the ideal body weight (using the upper limit of the midpoint range in the Metropolitan Tables for Life Insurance, 1983) x 100). Last observation carried forward was used for early terminated subjects.
Time Frame: Baseline to 24 months
Population: Intent to Treat Population - All subjects implanted with gastric band and signing informed consent.
Measure: Mean (Standard Deviation); unit: percent of excess weight at baseline
Arm/Group | Realize Adjustable Gastric Band-C
Number analyzed (Participants) | 231
percent of excess weight at baseline | 39.8 (25.12)
Statistical Analysis 1: Comparison: Realize Adjustable Gastric Band-C; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — One-sample t-test for change from baseline; Mean Difference (Final Values) = 39.8, 95% CI [36.6 to 43.1], Standard Deviation 25.12

2. Secondary Outcome: % Excess Weight Change From Baseline to 12 Months
Description: Percent excess weight change from baseline to 12 months was calculated as (the baseline weight minus the weight at 12 months) divided by the (baseline weight minus the ideal body weight (using the upper limit of the midpoint range in the Metropolitan Tables for Life Insurance, 1983) x 100). Last observation carried forward was used for early terminated subjects.
Time Frame: Baseline to 12 months
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: percent of excess weight at baseline
Arm/Group | Realize Adjustable Gastric Band-C
Number analyzed (Participants) | 231
percent of excess weight at baseline | 36.6 (19.79)
Statistical Analysis 1: Comparison: Realize Adjustable Gastric Band-C; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 36.6, 95% CI [34.0 to 39.2], Standard Deviation 19.79

3. Secondary Outcome: Change in Body Mass Index From Baseline to 24 Months
Description: Change in Body Mass Index from Baseline to 24 months with last observation carried forward. The calculation was performed as the Body Mass Index at 24 months minus the Body Mass Index at Baseline.
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: kilograms per meters squared
Arm/Group | Realize Adjustable Gastric Band-C
Number analyzed (Participants) | 231
kilograms per meters squared | -7.97 (5.233)
Statistical Analysis 1: Comparison: Realize Adjustable Gastric Band-C; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -7.97, 95% CI [-8.65 to -7.29], Standard Deviation 5.233

ADVERSE EVENTS:
Arm/Group | Realize Adjustable Gastric Band-C
Serious Adverse Events (participants affected / at risk) | 9/231
Other Adverse Events (participants affected / at risk) | 200/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Realize Adjustable Gastric Band-C (N=231)
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Device migration (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Medical device complication (Injury, poisoning and procedural complications) | 2
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 1
Oxygen saturation decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Realize Adjustable Gastric Band-C (N=231)
Abdominal pain (Gastrointestinal disorders) | 99
Vomiting (Gastrointestinal disorders) | 71
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 50
Dysphagia (Gastrointestinal disorders) | 48
Nausea (Gastrointestinal disorders) | 37
Procedural pain (Injury, poisoning and procedural complications) | 33
Constipation (Gastrointestinal disorders) | 15
Injection site pain (General disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed that the first publication of results should be made in conjunction with the presentation of a joint, multicenter publication of the results with the PIs from all sites contributing data, analyses, and comments. If this publication was not submitted within 12 months after conclusion of the Study at all sites, or after Sponsor confirmed there would be no multicenter Study publication, whichever is first, the PIs could have published the results from their individual sites.